CLINICAL TRIAL: NCT01649089
Title: Evaluation of Physical Function and Quality of Life (QOL) Before and After Non-Radical Surgical Therapy (Extra Fascial Hysterectomy or Cone Biopsy With Pelvic Lymphadenectomy) for Stage IA1 (LVSI+) and IA2-IB1 (≤ 2CM) Cervical Cancer
Brief Title: Studying the Physical Function and Quality of Life Before and After Surgery in Patients With Stage I Cervical Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GOG-0278; NCI-2012-01990 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000737208; GOG-0278 (Other: NRG Oncology); GOG-0278 (Other: DCP); GOG-0278 (Other: CTEP); U10CA101165 (NIH); U10CA180868 (NIH); UG1CA189867 (NIH)
Record Dates: First submitted 2012-07-21; First posted 2012-07-25 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Lymphedema; Stage IA1 Cervical Cancer AJCC v6 and v7; Stage IA2 Cervical Cancer AJCC v6 and v7; Stage IB1 Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Lymphedema | interventions — Conization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cone biopsy/lymphadenectomy or hysterectomy) (Experimental): Patients undergo cone biopsy and pelvic lymphadenectomy or simple hysterectomy and pelvic lymphadenectomy.
  Interventions: Procedure: Conization; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery; Procedure: Therapeutic Lymphadenectomy

INTERVENTIONS:
Procedure: Conization — Undergo cone biopsy
  Other Names: cone biopsy; Cone Biopsy of Cervix; Conization of Cervix; Conization of Uterine Cervix
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Therapeutic Conventional Surgery — Undergo hysterectomy
Procedure: Therapeutic Lymphadenectomy — Undergo lymphadenectomy

SUMMARY:
This clinical trial studies the physical function and quality-of-life before and after surgery in patients with stage I cervical cancer. Studying quality-of-life in patients undergoing surgery for cervical cancer may help determine the intermediate-term and long-term effects of surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the changes before and after non-radical surgical treatment (simple hysterectomy or cone biopsy [fertility preservation] and pelvic lymphadenectomy) on functional outcomes of bladder, bowel, and sexual function for stage IA1 (lymphatic vessel invasion positive [LVSI+]) and IA2-IB1 (=< 2 cm) carcinoma of the cervix.

II. To evaluate incidence and severity of lymphedema after non-radical surgery (simple hysterectomy or cone biopsy [fertility preservation] and pelvic lymphadenectomy) for stage IA1 (LVSI+) and IA2-IB1 (=< 2 cm) carcinoma of the cervix.

SECONDARY OBJECTIVES:

I. To investigate if non-radical surgery (simple hysterectomy or cone biopsy [fertility preservation] with pelvic lymphadenectomy) demonstrates greater physical function and less toxicity in comparison to historical data on radical surgery (radical hysterectomy or radical trachelectomy).

II. To evaluate incidence and severity of treatment-related adverse events, including surgical complications, among the entire cohort and by treatment type.

III. To evaluate changes in quality of life (QOL) (Functional Assessment of Cancer Therapy-Cervix [FACT-Cx]), cancer worries (Impact of Events Scale [IES]) and sexual (Female Sexual Function Index [FSFI])/reproductive concerns (RCS) among the entire cohort and by treatment type.

IV. To explore relationships (correlation, interaction, independence) between functional outcomes (i.e., bladder function, bowel function, sexual function), adverse events (including and surgical complication lymphedema [Gynecologic Cancer Lymphedema Questionnaire (GCLQ)]), cancer worry (IES), surgical complications, and overall quality of life (FACT-Cx).

V. To determine participants' intention for conception & fertility rates (Integrative Care for Fertility [ICF]) and assess the reproductive concerns (RCS) of women following cone biopsy and pelvic lymphadenectomy for stage IA1 (LVSI+) and IA2-IB1 (=< 2 cm) carcinoma of the cervix.

VI. To estimate the efficacy of non-radical surgery (simple hysterectomy or cone biopsy [fertility preservation] and pelvic lymphadenectomy) for stage IA1 (LVSI+) and IA2-IB1 (=< 2 cm) carcinoma of the cervix.

OUTLINE:

Patients undergo cone biopsy and pelvic lymphadenectomy or simple hysterectomy and pelvic lymphadenectomy.

Patients complete the FACT-Cx, the IES, the FSFI, the GCLQ, and the Patient Reported Outcomes Measurement Information System (PROMIS) questionnaires at baseline, 4-6 weeks after surgery, and then every 6 months for 3 years. Patients undergoing cone biopsy and pelvic lymphadenectomy also complete the ICF and RCS questionnaires.

After completion of study treatment, patients are followed up at 4-6 weeks, every 3 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must consent for the appropriate surgery
* Patients with a histologic diagnosis of squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma of the cervix, stage IA1 (lymph-vascular space invasion [LVSI]+), IA2, and IB1 (tumor size [maximum visible or palpable]) =< 2 cm), any grade
* All patients must have undergone a cone biopsy or loop electrosurgical excision procedure (LEEP); depth of invasion must be =< 10 mm
* Patients must have no evidence of metastasis on positron emission tomography (PET) scan or magnetic resonance imaging (MRI) or computed tomography (CT) scan of the pelvis and chest imaging
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patient must have Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2

Exclusion Criteria:

* Patients with stage IA1 disease who are LVSI negative
* Patients with stage IB1 with tumor size (maximum visible or palpable) > 2 cm
* Patients with >= stage IB2 disease
* Patients with clear cell or neuroendocrine cell types
* Patients with depth of invasion > 10 mm on first cone biopsy (or LEEP)
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2013-06-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in bladder and bowel function score based on supplemental bladder and bowel questions plus 4 items from the Functional Assessment of Cancer Therapy-Cervix (3 bladder and 1 bowel question) | Baseline to 3 years
  Analysis of variance methods with repeated measurements and a time component will initially be used to determine whether there are significant changes over time.
Change in sexual function and activity based on Female Sexual Function Index (19 items) score plus 2 Patient Reported Outcomes Measurement Information System screener items | Baseline to 3 years
  Analysis of variance methods with repeated measurements and a time component will initially be used to determine whether there are significant changes over time.
Lymphedema | Up to 3 years
  Based on Cancer Lymphedema Questionnaire score.
Maximum grade and duration of severe adverse events associated with bladder, bowel, and sexual dysfunction and lymphedema | Up to 3 years after non-radical surgical procedure
  Graded according to Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 will be used staring April 1, 2018).

SECONDARY OUTCOMES:
Maximum grade of treatment-related adverse events | Up to 30 days after surgical procedure
  Graded according to Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 will be used staring April 1, 2018).
Change in overall quality of life | Baseline to 3 years
  Will be assessed based on Functional Assessment of Cancer Therapy-Cervix (15 items) score. Analysis of variance methods with repeated measurements and a time component will initially be used to determine whether there are significant changes over time.
Change in cancer worries based on Impact of Events score | Baseline to 3 years
  Analysis of variance methods with repeated measurements and a time component will initially be used to determine whether there are significant changes over time.
Change in reproductive concerns based on reproductive concerns (14 items) score | Baseline to 3 years
  Analysis of variance methods with repeated measurements and a time component will initially be used to determine whether there are significant changes over time.
Site of first recurrence | Up to 3 years
  Classified as either local (pelvis regions, including vaginal) or distant (abdomen, lung, bone, brain, and other).
Recurrence-free survival | Up to 3 years
  Product-limit estimates according to the method of Kaplan and Meier will be used to estimate recurrence-free survival. In addition, Cox proportional hazard regression will be employed to evaluate relative risk (hazard ratio) adjusting for known prognostic factors. Trellis plots will be used to display point estimates of hazard ratio and respective 95% confidence intervals from subgroup analyses. Local recurrence will be summarized using frequency tables and plot of cumulative incidence of local recurrence over time.
Overall survival | Up to 3 years
  Product-limit estimates according to the method of Kaplan and Meier will be used to estimate overall survival. In addition, cox proportional hazard regression will be employed to evaluate relative risk (hazard ratio) adjusting for known prognostic factors. Trellis plots will be used to display point estimates of hazard ratio and respective 95% confidence intervals from subgroup analyses. Gompertz hazard regression will also be employed to evaluate relative risk (hazard ratio) and cure rates, adjusting for known prognostics factors.

CONTACTS AND LOCATIONS:
Overall Officials: Allan L Covens, Principal Investigator — NRG Oncology
Locations (185):
- United States (174):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- South Korea (10):
  - Samsung Medical Center, Seoul, Korea
  - Catholic University of Korea-Seoul Saint Mary's Hospital, Seoul, Korea
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System-Severance Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Korea Cancer Center Hospital, Seoul

REFERENCES:
- [Derived] Boisen M, Guido R. Emerging Treatment Options for Cervical Dysplasia and Early Cervical Cancer. Clin Obstet Gynecol. 2023 Sep 1;66(3):500-515. doi: 10.1097/GRF.0000000000000790. Epub 2023 Jul 25. PMID 37650664